CLINICAL TRIAL: NCT02020135
Title: An Open-label Treatment Extension of PSMA ADC in Subjects With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: An Open-label Extension Study of PSMA ADC 2301 in mCRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSMA ADC 2301EXT
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PSMA ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: PSMA ADC (Experimental): Subjects started the extension study at the same dose received upon completion of the core PSMA ADC 2301 study. Each Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) dose was administered as an IV infusion over approximately 60 minutes once every three weeks (Q3W) for up to eight doses, unless a dose delay or dose reduction was required.
  Interventions: Drug: PSMA ADC

INTERVENTIONS:
Drug: PSMA ADC — Upon recommendation from the PI and after Sponsor approval, a subject benefiting from treatment could have received up to eight additional doses Q3W. Subjects were weighed prior to each cycle and dosing was calculated on a mg/kg basis prior to each dose, with a maximum weight of 100 kg for dosing calculations.

SUMMARY:
PSMA ADC 2301EXT is an open-label study to further assess the anti-tumor activity as measured by radiographic imaging and biomarkers, safety and tolerability of Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) in subjects with mCRPC. Subjects who have participated in the PSMA ADC 2301 study and who, in the opinion of the Principal Investigator are likely to benefit from continued treatment with PSMA ADC are eligible for the PSMA ADC 2301 extension study. Subjects who are benefiting from treatment may be able to receive up to an additional eight to sixteen doses (every 3 weeks) of PSMA ADC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed the PSMA ADC 2301 study and who, in the opinion of the investigator, are likely to benefit from continued treatment with PSMA ADC
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
3. If chemically castrated, subjects must agree to stay on androgen-deprivation therapy for the duration of the study
4. If applicable, men must agree to commit to the use of a medically acceptable method of birth control (e.g., spermicide in conjunction with a barrier such as a condom) or sexual abstinence for the duration of the study, including 30 days after the last dose of study drug

Exclusion Criteria:

1. An acute infection requiring ongoing antibiotic therapy (e.g., UTI, indwelling catheter or other potential site(s) of infection)
2. History of significant hypersensitivity reactions to PSMA ADC or any of its components, or to any prior investigational or approved monoclonal antibodies (mAbs), immunoglobulin (Ig) fusion proteins (e.g., circulating neutralizing antibodies), or ADC
3. Clinically significant cardiac disease or severe debilitating pulmonary disease
4. Any recent or ongoing medical condition that may interfere with a subject's participation or compliance with the study or evaluation of PSMA ADC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Wong, PhD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Tucson, Arizona
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Las Vegas, Nevada
  - Stony Brook, New York
  - Myrtle Beach, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PSMA ADC: Subjects started the extension study at the same dose received upon completion of the core PSMA ADC 2301 study. Each PSMA ADC dose was administered as an IV infusion over approximately 60 minutes once every three weeks (Q3W) for up to eight doses, unless a dose delay or dose reduction was required.
  PSMA ADC: Upon recommendation from the PI and after Sponsor approval, a subject benefitting from treatment could have received up to eight additional doses Q3W. Subjects were weighed prior to each cycle and dosing was calculated on a mg/kg basis prior to each dose, with a maximum weight of 100 kg for dosing calculations.
Period: Overall Study
Arm/Group | Arm 1: PSMA ADC
Started | 9
Completed | 0
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- PSMA ADC Chemotherapy-experienced; PSMA ADC Chemotherapy-naive: Subjects started the extension study at the same dose received upon completion of the core PSMA ADC 2301 study. Each Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) dose was administered as an IV infusion over approximately 60 minutes once every three weeks (Q3W) for up to eight doses, unless a dose delay or dose reduction was required.
  PSMA ADC: Upon recommendation from the PI and after Sponsor approval, a subject benefitting from treatment could have received up to eight additional doses Q3W. Subjects were weighed prior to each cycle and dosing was calculated on a mg/kg basis prior to each dose, with a maximum weight of 100 kg for dosing calculations.
- Total: Total of all reporting groups
Arm/Group | PSMA ADC Chemotherapy-experienced | PSMA ADC Chemotherapy-naive | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Full Range); unit: years] | 73.2 [66 to 81] | 77.3 [70 to 84] | 74.6 [66 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 3 | 9
Prostate specific antigen (PSA) [Mean (Standard Deviation); unit: ug/mL] | 1446.3 (2209.9) | 91.3 (125.8) | 994.6 (1874.9)
PSA [Median (Full Range); unit: ug/mL] | 442.2 [107.9 to 5781.1] | 32.1 [6.0 to 235.8] | 221.2 [6.0 to 5781.1]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total Serum PSA Response
Description: Total serum PSA (prostate-specific antigen) was measured at baseline and had at least one post-baseline assessment. PSA response was examined at two levels: at least 30% decrease or at least 50% decrease in serum PSA. Response was assessed as the maximum decrease over the extension study. Response was defined as any decrease from baseline of at least 30% or 50%.
Time Frame: 25 Weeks
Population: Both groups must also have received and progressed on abiraterone acetate and/or enzalutamide prior to the study (once these agents were commercially available for use). The population examined was those subjects with a PSA baseline value and at least one post-baseline value.
Measure: Number; unit: % of responders
Groups:
- PSMA ADC Chemotherapy-experienced: The chemotherapy-experienced group was comprised of 6 subjects who must have received at least one taxane-containing chemotherapy regimen (e.g., docetaxel, cabazitaxel) prior to the study (more than two cytotoxic chemotherapy regimens required sponsor approval for study participation).
  Subjects started the extension study at the same dose received upon completion of the core PSMA ADC 2301 study. Each PSMA ADC dose was administered as an IV infusion over approximately 60 minutes once every three weeks (Q3W) for up to eight doses, unless a dose delay or dose reduction was required.
- PSMA ADC Chemotherapy-naive: The chemotherapy-naïve group was comprised of 3 subjects who were cytotoxic chemotherapy-naïve. Chemotherapy-naïve subjects must have received and progressed on Radium-223 (following its approval by FDA), or have been ineligible for it, refused it, had an intolerance to it, or did not have access to it.
  Subjects started the extension study at the same dose received upon completion of the core PSMA ADC 2301 study. Each PSMA ADC dose was administered as an IV infusion over approximately 60 minutes once every three weeks (Q3W) for up to eight doses, unless a dose delay or dose reduction was required.
Arm/Group | PSMA ADC Chemotherapy-experienced | PSMA ADC Chemotherapy-naive
Number analyzed (Participants) | 6 | 3
% of responders
  >30% Decrease in PSA | 67 | 33
  >50% Decrease in PSA | 33 | 0

2. Primary Outcome: CTC Response
Description: Circulating tumor cells (CTC) response was measured at baseline and had at least one post-baseline assessment. Response was assessed as the maximum decrease over the extension study. Response was defined as any decrease from baseline of at least 50%.
Time Frame: 25 weeks
Population: Both groups must also have received and progressed on abiraterone acetate and/or enzalutamide prior to the study (once these agents were commercially available for use). The population examined was those subjects with a CTC baseline value and at least one post-baseline value.
Measure: Number; unit: % of responders
Arm/Group | PSMA ADC Chemotherapy-experienced | PSMA ADC Chemotherapy-naive
Number analyzed (Participants) | 5 | 2
% of responders | 100 | 50

3. Primary Outcome: Overall Radiologic Response
Description: Overall radiologic response was measured at baseline and post-baseline. Imaging techniques used at screening were used throughout the study. The preferred imaging techniques include: bone scan, contrast enhanced CT of chest, contrast enhanced CT of pelvis, and contrast enhanced CT of upper & lower abdomen. Best overall radiologic response (confirmed), target and non-target lesions, was defined as responses in bone, visceral or nodal metastases according to the Modified Response Evaluation Criteria (RECIST 1.1). The best overall radiologic response is the best response recorded from the start of the treatment until disease progression/recurrence (taking, as reference for progressive disease, the smallest measurements recorded since the treatment started). The subject's best response assignment depended on the achievement of both measurement and confirmation criteria.
Time Frame: 25 weeks
Population: Both groups must also have received and progressed on abiraterone acetate and/or enzalutamide prior to the study (once these agents were commercially available for use). All subjects (n=9) enrolled in 2301EXT were evaluated.
Measure: Number; unit: % of subjects
Arm/Group | PSMA ADC Chemotherapy-experienced | PSMA ADC Chemotherapy-naive
Number analyzed (Participants) | 6 | 3
% of subjects
  Partial response | 17 | 0
  Stable disease | 83 | 100

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | PSMA ADC Chemotherapy-experienced | PSMA ADC Chemotherapy-naive
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PSMA ADC Chemotherapy-experienced (N=6) | PSMA ADC Chemotherapy-naive (N=3)
Tachycardia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PSMA ADC Chemotherapy-experienced (N=6) | PSMA ADC Chemotherapy-naive (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Arrythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Gait disturbance (General disorders) | 1 | 1
Gravitational edema (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Peripheral edema (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Peripheral neuropathy (Nervous system disorders) | 6 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No